CLINICAL TRIAL: NCT00964704
Title: A Single Arm, Open-label Study to Evaluate the Efficacy on Tumor Response and the Safety of Bevacizumab and Trastuzumab Combination and Sequential Capecitabine in Patients With HER2 +Ive Locally Recurrent or Metastatic Breast Cancer After Early Relapse to Adjuvant Trastuzumab-containing Therapy
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With Avastin (Bevacizumab) and Sequential Xeloda (Capecitabine) or Docetaxel in Patients With HER2-Positive Locally Recurrent or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients have been recruited therefore study has been cancelled
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22056; 2008-007495-20
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Capecitabine; Docetaxel; Trastuzumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: docetaxel; Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv every 3 weeks
Drug: capecitabine [Xeloda] — added at time of disease-progression, 1000mg/m2 bid po days 1-14 of every 3-week cycle
Drug: docetaxel — background therapy at time of disease progression, 100mg/m2 iv every 3 weeks
Drug: trastuzumab [Herceptin] — 8mg/kg iv on day 1 of the first 3-week cycle, followed by 6mg/kg every 3 weeks

SUMMARY:
This single arm, open-label study will evaluate the safety and efficacy of Herceptin in combination with Avastin and sequential Xeloda in patients with locally recurrent or metastatic HER2-positive breast cancer after early relapse on adjuvant Herceptin therapy. Patients will receive Herceptin at a loading dose of 8mg/kg iv followed by 6mg/kg iv every three weeks, and Avastin 15mg/kg every 3 weeks. At first sign of disease progression Xeloda 1000mg/m2 bid po will be added on days 1-14 of each cycle, or docetaxel (100mg/m2 iv every 3 weeks) if Xeloda is not indicated for a patient. Anticipated time on study treatment is until disease-progression on second line treatment and target sample size is <100.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, age >/=18 years
* locally recurrent or metastatic HER2-positive breast cancer
* disease progression during or up to 12 months after prior adjuvant therapy with trastuzumab
* LVEF >/=55% at baseline

Exclusion Criteria:

* prior treatment with bevacizumab or capecitabine
* anthracyclines in prior adjuvant or neoadjuvant treatment exceeding cumulative dose of 360mg/m2 for doxorubicin and 720mg/kg for epirubicin
* chronic daily treatment with corticosteroids (>10mg/day methylprednisolone equivalent; excluding inhaled corticosteroids), or aspirin (>325mg/day), or clopidogrel (>75mg/day)
* clinically significant cardiac disease, or cardiac toxicity during previous trastuzumab therapy
* evidence of spinal cord compression or CNS metastasis
* history of other malignancy, unless disease-free for >/=5 years or treated curatively for carcinoma in situ of the cervix or non-melanomatous skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival on second-line treatment | event-driven, tumour assessments every 6 weeks for 24 weeks, every 12 weeks thereafter

SECONDARY OUTCOMES:
Safety and tolerability: AEs, laboratory parameters, LVEF | throughout study, laboratory parameters every 3 weeks, LVEF every 12 weeks
Overall Response Rate, Best Overall Response, Duration of Response, Progression-free Survival (first-line), Overall Survival | event-driven, tumour assessment every 6 weeks for 24 weeks, every 12 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche